CLINICAL TRIAL: NCT02402426
Title: Brain Health Registry - Online Registry for Brain Research
Brief Title: Brain Health Registry: An Online Registry to Identify and Assess Subjects for Brain Research
Acronym: BHR
Status: Enrolling by invitation | Type: Observational
Sponsor: University of California, San Francisco (Other)
Responsible Party: Sponsor
Other Study IDs: 12-09628
Record Dates: First submitted 2013-08-01; First posted 2015-03-30 (Estimated); Last update posted 2026-01-13 (Actual); Status verified 2026-01

CONDITIONS: Healthy; Neurodegenerative Disease
Keywords: Brain Health; Brain Research; Alzheimer's Disease; Neurodegenerative Disease; Parkinson's Disease; Dementia; Stroke; PTSD; Multiple Sclerosis
MeSH Terms: conditions — Neurodegenerative Diseases; Alzheimer Disease; Parkinson Disease; Dementia; Stroke; Stress Disorders, Post-Traumatic; Multiple Sclerosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 10 Years
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The overall goal of this project is to identify, assess and longitudinally monitor subjects who are interested in participating in brain research. Participants will enroll through the website, BrainHealthRegistry.org, and provide informed consent prior to any study activities. The website will collect a variety of information, including participants' overall health, memory complaints, family history of dementia and Alzheimer's disease (AD), mood status, sleep, diet, and exercise-all through self-reported online questionnaires. Participants will also be ask to take online cognitive tests, and to return to the website at regular intervals, to complete follow-up questionnaires and neuropsychological assessments. Everyone over the age of 18 is welcome to participate. To join the Brain Health Registry, please visit www.BrainHealthRegistry.org.

DETAILED DESCRIPTION:
Through advertisement and community outreach, potential participants will be directed to the website, BrainHealthRegistry.org. The overall goal of this project is to identify, assess and longitudinally monitor subjects who are interested in participating in brain research. Participants will enroll through the website, BrainHealthRegistry.org, and provide informed consent prior to any study activities.

The website will include:

1. Information about the Brain Health Registry (who is eligible to participate, the goals of the project and other relevant information about investigators and sponsors involved in the Initiative)
2. Frequently Asked Questions (FAQs) such as "How will my information be used?", "How will patient information be safeguarded?", "What information will be requested?", "How much time will be required for registration and testing?" will be addressed for participants.
3. General information about Alzheimer's disease and other neurodegenerative diseases discussed in lay terms Links to sites that may be of interest to participants
4. Login to our secure Registry website

The Registry will be a large, online database of volunteers who are interested in participating in neuroscience research. While anyone over the age of 18 is welcome to join the Registry, the intent is to concentrate all efforts on enrolling participants age 55 years and older. It will consist of online tools and databases, which are HIPAA-compliant and secure.

1. Participants will access the Registry by going to the BHR website, BrainHealthRegistry.org
2. Participants will provide their email address and create an account and user name with the Registry
3. The Registry will send an automatic email to the participant to verify their email address
4. Participants will read the online Information Sheet and will be asked to provide their consent by clicking either "I consent" or "I decline." Participants who decline to participate in the Registry will be automatically directed out of the Registry website
5. Participants who give their consent will be permitted to continue through the registration process, which includes completing a battery of questionnaires designed to obtain a general understanding of participants health, medical history wellbeing
6. In addition to questionnaires, participants will be able to complete online cognitive assessments.
7. Participants will given the option to elect a Caregiver and/or Study Partner (CASP) to enrich their study profile.
8. Participants may be referred to other research studies and/or clinical trials

ELIGIBILITY:
Inclusion Criteria:

* Anyone over the age of 18 is welcome to join the Registry

Exclusion Criteria:

* N/A

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The Registry is a large, online database of volunteers who would like to participate in clinical trials and research. Anyone over the age of 18 is welcome to join the Registry, and the intent is to concentrate all efforts on enrolling participants age 55 years and older.
Sampling Method: Non-Probability Sample
Enrollment: 200000 (Estimated)
Dates: Start 2013-09; Primary Completion 2030-09 (Estimated); Study Completion 2030-09 (Estimated)

PRIMARY OUTCOMES:
Alzheimer's Disease | 10 years
  The overall goal of The Brain Health Registry is to facilitate and accelerate treatments for diseases which affect the brain.

SECONDARY OUTCOMES:
Neurodegenerative Diseases | 10 years
  The main goal of this project is to promote healthy brain aging through the prevention of Alzheimer's disease and other neurodegenerative diseases such as Parkinson's disease, depression, stroke and other conditions that affect brain function in older adults. Our broader goal is to develop an innovative model for subject recruitment and clinical trials of treatments for brain disorders across the age spectrum.

CONTACTS AND LOCATIONS:
Overall Officials: Michael Weiner, MD, Principal Investigator — University of California, San Francisco
Locations (1):
- BrainHealthRegistry.org, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Brain Health Registry: How it works; Join — http://www.brainhealthregistry.org/